CLINICAL TRIAL: NCT06450418
Title: Digital App for Speech & Health Monitoring in Neurodegenerative Disorders
Brief Title: Digital App for Speech & Health Monitoring
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC24003
Record Dates: First submitted 2024-02-09; First posted 2024-06-10 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Dementia; Motor Neuron Disease; Multiple Sclerosis; Parkinson Disease
MeSH Terms: conditions — Dementia; Motor Neuron Disease; Multiple Sclerosis; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Participants can additionally and optionally consent for blood samples to be obtained during the study. These samples will be collected and stored with the intention of exploring emerging blood-based biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Carers/Realtives/ Healthy - No Diagnosis of a Neurodegenerative Disorder
- Motor Neuron Disease
- Multiple Sclerosis
- Dementia
- Parkinson's Disease

SUMMARY:
Many people living with neurodegenerative conditions like dementia, motor neuron disease (MND), multiple sclerosis (MS), and Parkinson's disease (PD), suffer from speech problems. Using common digital technologies such as smartphone apps, the investigators can record and analyse speech in detail to provide new information for people living with these conditions, researchers, and healthcare professionals. This study will investigate the use of these digital speech recordings to help diagnose and monitor these conditions.

To take part, participants will have either a diagnosis of dementia, motor neuron disease, Parkinson's disease or Multiple Sclerosis, OR they will have no diagnosis of a neurological condition. Researchers will compare people with a diagnosis of a Neurological condition to those without.

DETAILED DESCRIPTION:
This project aims to create novel speech-based solutions for: 1) Early detection, 2) Monitoring and 3) Stratification of neurodegenerative disorders including dementia, motor neuron disease (MND), Parkinson's disease (PD), and multiple sclerosis(MS). The investigators will develop and validate proof of concept and early-stage algorithms derived from acoustic data, which will be scaled and tested in deeply-phenotyped population.

2.2 Objectives Primary Objectives

1. To deploy and iterate a digital platform, co-produced with people living with neurodegenerative disorders, for acquisition of speech data from well characterised cohorts of people living with neurodegenerative disorders (dementia, motor neuron disease, multiple sclerosis, Parkinson's disease), and a healthy control cohort (comprising relatives/carers and volunteers without a neurological diagnosis), linked to our highly curated clinical registries at the Anne Rowling Regenerative Neurology Clinic.
2. To collect a large body of acoustic speech data from well characterised cohorts of people living with neurodegenerative disorders (dementia, MND/ALS, multiple sclerosis, Parkinson's disease), and a healthy control cohort (comprising relatives/carers and volunteers without a neurological diagnosis), linked to highly curated clinical registries.
3. To apply machine learning approaches directly to acoustic and linguistic signals from voices from people with dementia, MND, MS, Parkinson's, and healthy controls (comprising relatives/carers and volunteers without a neurological diagnosis), and to characterise prosodic patterns (rhythm, intonation, and fluency) without explicit reference to the text which is spoken, providing powerful cues about the health of the speaker.
4. Compare speech based digital outcome measures to current clinical standards to characterise and validate their clinimetric properties.

Secondary Objectives

1. Assess the feasibility and acceptability of a digital outcome measure platform in people living with neurodegenerative conditions, for use in clinical care and research.
2. To create a repository of well characterised acoustic voice samples for open access sharing/collaboration with research and industry partners.

ELIGIBILITY:
Inclusion Criteria - Any one of the following:

* A person with a diagnosis of Motor Neuron Disease, Dementia, Multiple Sclerosis, or Parkinson's Disease.
* A relative or carer of the above who does not report to have a neurological condition.
* A healthy volunteer who does not report to have a neurological condition.

Exclusion Criteria:

* Age <16 years
* Significant and uncorrected visual or hearing impairment (precluding use of the App).
* Lack capacity to consent to project due to cognitive impairment (precluding understanding of the study and use of the App).

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with Neurodegenerative Disorders and their relatives or carers without a diagnosis of a Neurodegenerative disorder.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measures | 24 months
  Area under the curve (AUC) of the receiver operating characteristic (ROC) curve for each of the 4 binary classifiers distinguishing between a disease-positive group and a healthy control group.

SECONDARY OUTCOMES:
Secondary outcome measure | 24 months
  Sensitivity, specificity, positive and negative predictive values for each of the 4 binary classifiers distinguishing between a disease-positive group and a healthy control group.
Secondary outcome measure | 24 months
  Mean squared error of 4 regression models making predictions of condition-specific clinical rating scores (ACE-III, ALSFRS-R, EDSS, MDS-UPDRS)

CONTACTS AND LOCATIONS:
Overall Officials: Suvankar Pal, Prof, Principal Investigator — University of Edinburgh
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tam J, Weaver C, Ihenacho A, Newton J, Virgo B, Barrett S, Neale J, Perry D, Smith A, Chandran S, Watts O, Pal S; DASH Consortium. Digital App for Speech and Health Monitoring Study (DASH): protocol for a prospective longitudinal case-control observational study for developing speech datasets in neurodegenerative disorders and dementia. BMJ Open. 2025 Dec 5;15(12):e100222. doi: 10.1136/bmjopen-2025-100222. PMID 41360452